CLINICAL TRIAL: NCT05885022
Title: Feasibility Clinical Evaluation of the Calibreye System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Myra Vision Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFP-101, CFP-103
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Glaucoma Drainage Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Investigational Device Arm (Experimental): Subjects will receive a Calibreye glaucoma device (permanent implant)
  Interventions: Device: Calibreye System

INTERVENTIONS:
Device: Calibreye System — Implantation of a glaucoma device to reduce intraocular pressure
  Other Names: Glaucoma device, Glaucoma implant, Aqueous Shunt

SUMMARY:
To evaluate the safety and feasibility of the Calibreye System in patients with open angle glaucoma.

DETAILED DESCRIPTION:
This is a prospective, nonrandomized, open-label feasibility clinical trial, to evaluate the surgical procedure, safety and effectiveness of the Calibreye System in reducing intraocular pressure in subjects with open angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Open angle, pseudoexfoliative or pigmentary glaucoma
* IOP at preoperative visit of ≥ 18mmHg and ≤ 45mmHg
* Visual field mean deviation score of -3dB or worse
* Area of healthy, free and mobile conjunctiva in the target quadrant
* Shaffer angle grade ≥ 3 in the target quadrant

Exclusion Criteria:

* Angle closure glaucoma
* Congenital, neovascular or other secondary glaucomas
* Previous intraocular surgery (with the exception of laser trabeculoplasty or uncomplicated phacoemulsification with IOL occurring > 3 months prior to the preoperative visit)
* Previous glaucoma shunt/valve in the target quadrant
* Clinically significant inflammation or infection in the study eye within 30 days prior to the preoperative visit
* History of corneal surgery, corneal opacities or corneal disease
* Active diabetic retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure | 12 Months
  Percent change in IOP from baseline to the 12-month visit
Adverse Events | 12 Months
  Number and percentage of subjects having any adverse event

SECONDARY OUTCOMES:
Glaucoma Medication Usage | 12 Months
  Change in number of medications used compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Keith Barton, MD, Study Chair — Moorfields Eye Hospital NHS Foundation Trust
Locations (4):
- Dr. Agarwal's Eye Hospital Ltd., Chennai, India
- Mexico (2):
  - Centro Oftalmologico de Chihuahua, Chihuahua City
  - Oftalmología Láser de Puebla S.C., Puebla City
- Panama Eye Center, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No